CLINICAL TRIAL: NCT00082979
Title: Evaluation of the Role of Duct Endoscopy in the Assessment of Cellular Atypia Within Breast Duct Fluid in High-Risk Women Carrying BRCA1/2 or p53 Gene Mutations
Brief Title: Duct Endoscopy in Assessing Cellular Atypia in the Breast Duct Fluid of Women With a Genetic Risk for Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Diagnostic
Other Study IDs: CDR0000361751; RMNHS-2282; EU-20351
Record Dates: First submitted 2004-05-14; First posted 2004-05-17 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2005-12

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cytogenetic Analysis; Immunohistochemistry

INTERVENTIONS:
Genetic: cytogenetic analysis
Genetic: proteomic profiling
Other: cytology specimen collection procedure
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Procedure: breast duct lavage

SUMMARY:
RATIONALE: Diagnostic procedures, such as breast duct endoscopy, may improve the ability to detect breast cancer earlier and plan more effective treatment.

PURPOSE: This phase II trial is studying how well breast duct endoscopy works in assessing cellular atypia (abnormal cells) in the breast ducts of women with a genetic risk for breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Correlate cell yield and morphology findings from ductal lavage with duct endoscopy findings and any subsequent surgical pathology findings in high-risk women with BRCA1, BRCA2, or p53 gene mutations who have cellular atypia.
* Determine the prevalence of occult breast cancer in patients with cellular atypia undergoing duct endoscopy.

Secondary

* Determine patient acceptance of duct endoscopy.
* Perform immunohistochemical analysis (including estrogen receptor, progesterone receptor, HER2-neu receptor, epidermal growth factor receptor, p53, and proliferation marker expression) for markers potentially associated with breast cancer in these patients.
* Determine potential molecular markers of malignancy by gene methylation, gene expression, and proteomics in these patients.

OUTLINE: Patients undergo nipple aspiration to identify productive ducts and collect fluid for tumor marker assessment followed by ductal lavage over 15 minutes. Patients undergo duct endoscopy over approximately 30 minutes under local anesthesia. If no abnormality is found, duct endoscopy is repeated in 6 months. If the repeat duct endoscopy is normal, patients continue to undergo nipple aspiration or ductal lavage as specified in protocols RMNHS-2242 and RMNHS-2269. If an abnormality is found during either the initial or repeat duct endoscopy, patients may undergo further assessment comprising imaging or biopsy and/or appropriate surgical intervention.

Fluid is analyzed for tumor markers by immunohistochemistry. Candidate genes are analyzed by gene methylation studies, gene expression arrays, and proteomic analysis.

Patients are followed for at least 5 years.

PROJECTED ACCRUAL: A total of 45-60 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of cellular atypia in nipple aspirate or ductal lavage fluid
* Enrollment on RMNHS-2242 or RMNHS-2269 required
* No inflammatory breast cancer
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 to 64

Sex

* Female

Menopausal Status

* Any status

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* No prior allergy to eutectic mixture of local anesthetics (EMLA®) cream or lidocaine
* No severe illness that would preclude study participation
* No mental illness or handicap that would preclude study compliance
* No active infection or inflammation in the breast being studied
* No nursing within the past 12 months
* Not pregnant
* Not unconscious

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* No prior tamoxifen

Radiotherapy

* Not specified

Surgery

* No prior subareolar surgery (e.g., papilloma resections, biopsies, or fine needle aspirations) or any other surgery that may disrupt the ductal systems within 2 cm of the nipple

  * Biopsies and fine needle aspirations > 2 cm from the nipple are allowed
* No prior breast implantation on proposed lavage side

Other

* No prior chemopreventative agents

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2003-10

PRIMARY OUTCOMES:
Comparison of cell yields and morphology from ductal lavage vs the ductal anatomy visualized at duct endoscopy
Prevalence of occult pathology (malignant and benign) as assessed by duct endoscopy on intraduct sampling
Sensitivity and specificity of ductal lavage to duct endoscopy in detecting atypia or malignancy
Comparison of cell yields vs final surgical pathology

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Gui, MD, MS, FRCS(Edin), FRCS(Eng) — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden - London, London, England, United Kingdom